CLINICAL TRIAL: NCT05016440
Title: Lisinopril To Reduce Microalbuminuria In Postpartum Preeclamptic Women. A Role For Renal Protection?
Brief Title: Lisinopril for Renal Protection in Postpartum Preeclamptic Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Lisinopril-Renal Protection
Record Dates: First submitted 2014-08-20; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Microalbuminuria; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Lisinopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lisinopril (Active Comparator): 10mg Lisinopril tablets
  Interventions: Drug: Lisinopril
- Sugar pill (Placebo Comparator): sugar pill
  Interventions: Drug: Lisinopril

INTERVENTIONS:
Drug: Lisinopril — 10mg Lisinopril daily for 6-8 weeks postpartum

SUMMARY:
There may be a role for Lisinopril in improving renal protection in post-partum women who had preeclampsia during pregnancy. The aim of this study is to determine whether routine initiation of Lisinopril after delivery, in women who had preeclampsia while they were pregnant, can control high blood pressure and improve kidney function.

DETAILED DESCRIPTION:
This study is being done to determine the effects (good or bad) of Lisinopril (high blood pressure medication) in controlling high blood pressure and improving kidney function for women after delivery who had preeclampsia while they were pregnant .Preeclampsia is a condition that can occur during pregnancy, up to 6 weeks post partum, where the mother's blood pressure is high and protein is present in the urine. This can be dangerous for both the mother and fetus. Although the blood pressure usually returns to normal after delivery, elevated pressures may continue. Normally medication is given when you continue to have high blood pressure after delivery. High blood pressure can cause damage to the kidneys. Lisinopril is a medication that can be used to treat high blood pressure after delivery. Lisinopril offers kidney protection in patients diagnosed with diabetes. We currently do not know if lisinopril can offer the same kidney protection in women diagnosed with preeclampsia. Considering that 10% of all pregnant women develop preeclampsia, the number of women who may eventually develop end stage kidney disease is relatively large and any relatively safe and easy means to prevent this disease would be beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 to 50 yrs of age with mild or severe preeclampsia diagnosed using criteria (listed below) set forth by the American College of Obstetrics and Gynecology (ACOG) Criteria. (Note; women who become eclamptic will be included in the study.)

  * Blood Pressure of 140 mmHg systolic or greater or 90 mmHg diastolic or higher that occurs after 20 weeks' gestational age in a woman with previously normal blood pressure
  * Proteinuria defined as 0.3 g protein or higher in a 24 hour urine specimen.
  * Preeclampsia was considered severe when any of the following were present:

    1. Blood pressure of 160 mmHg systolic of higher or 110 mg Hg diastolic or higher on two occasions at least 6 hours apart while the patient is on bed rest
    2. Proteinuria of 5 grams of higher in a 24-hour urine specimen of 3+ or greater on two random urine samples collected at least 4 hours apart
    3. Oliguria of less than 500cc in 24 hours
    4. Cerebral of visual disturbances
    5. Pulmonary edema or cyanosis
    6. Epigastric or right upper quadrant pain
    7. Impaired liver function, thrombocytopenia
    8. Fetal growth restriction.

Exclusion Criteria:

* Women with:

  * Prior hypersensitivity (allergic reaction) to Lisinopril or ACE Inhibitors
  * Pre-gestational chronic hypertension
  * Pre-gestational diabetes
  * Rheumatologic disorders (i.e., systemic lupus erythematosus, scleroderma)
  * Multiple gestations for present pregnancy
  * Patients who declined birth control postpartum
  * Patient who has been on an Ace-inhibitor within 6 months prior to pregnancy
  * Cardiac problems like; Aortic stenosis or Hypertrophic cardiomyopathy
  * Severe kidney disease
  * Myocardial infarction within the past 6 months
  * Taking any of the prohibited medications listed in section VI
  * Breast feeding
  * Prisoners will not be included in the study due to difficulty in tracking their pregnancy care being provided at the prison centers

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09 (Estimated); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Albumin Excretion Rate in mg/mmol | Change is being assessed within 24 hours of delivery and 6-8 weeks postpartum
  Prior to discharge from the hospital, either during the woman's labor progress or immediately post delivery, a catheterized urine specimen will be obtained and sent to the lab for an Albumin-Creatinine Ratio (ACR) by a nurse. Following discharge, the woman will be seen 6-8 weeks postpartum for her routine postpartum visit. If the woman reports vaginal spotting or bleeding a straight catheter urine specimen will be obtained, otherwise a clean catch specimen may be obtained, and sent for lab assessment of Albumin-Creatinine Ratio (ACR). This collection of a urine specimen is standard of care for our pregnant and postpartum patients. Prior to hospital discharge, she will also be instructed to collect a 24 hour urine specimen collection, the day before her 6-8 week postpartum visit and bring it with her to this visit. When analyzed, this second 24 hour urine specimen will be assessed for both albumin concentration and albumin/creatinine ratio (Albumin Excretion Rate).

CONTACTS AND LOCATIONS:
Overall Officials: James Hill, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States